CLINICAL TRIAL: NCT03839888
Title: Short Term Refractive and Ocular Parameter Changes After Topical Atropine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BuddhistTCGHTaipei2
Record Dates: First submitted 2019-02-10; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Myopia, Left Eye
Keywords: atropine; cycloplegia; refraction; axial length; anterior chamber depth
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 0.125% atropine group (Experimental): patients used the 0.125 % atropine eyedrop every night before sleep for 7 days
  Interventions: Drug: 0.125% Atropine

INTERVENTIONS:
Drug: 0.125% Atropine — patients used 0.125% atropine eyedrop per night before sleep for 7 days.

SUMMARY:
In order we had designed a prospective clinical trial. Spherical equivalent refractive error (SER), axial length (AL), mean keratometric value (Mean-K), anterior chamber depth (ACD), and intraocular pressure (IOP) were measured at baseline and one week after topical use of 0.125% atropine. Postcycloplegic changes of refractive error and ocular parameters were evaluated, and their correlations were analyzed with multiple linear regression models.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had an SER of -0.5 diopters or less in their eyes.

Exclusion Criteria:

* Patients who had already been undergoing cycloplegic treatment for myopia before.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
SER | change from SER at 7 days
  Spherical equivalent refractive error

SECONDARY OUTCOMES:
AL | change from AL at 7 days
  Axial length
ACD | change from ACD at 7 days
  anterior chamber depth
IOP | change from IOP at 7 days
  intraocular pressure

REFERENCES:
- [Derived] Ho MC, Hsieh YT, Shen EP, Hsu WC, Cheng HC. Short-term refractive and ocular parameter changes after topical atropine. Taiwan J Ophthalmol. 2019 Feb 20;10(2):111-115. doi: 10.4103/tjo.tjo_110_18. eCollection 2020 Apr-Jun. PMID 32874839